CLINICAL TRIAL: NCT05395715
Title: Conditioning Electrical Stimulation Enhances Recovery Following Surgery for Severe Cubital Tunnel Syndrome: A Double-Blind Randomized Controlled Trial
Brief Title: Conditioning Electrical Stimulation to Improve Outcomes in Cubital Tunnel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CuTS CES
Record Dates: First submitted 2022-04-18; First posted 2022-05-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cubital Tunnel Syndrome; Electrical Stimulation
Keywords: Cubital tunnel syndrome; Nerve regeneration; Electrical stimulation; Functional outcomes; Randomized control trial; Surgery; Peripheral nerve regeneration
MeSH Terms: conditions — Cubital Tunnel Syndrome | interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Control patients will receive cubital tunnel surgery and sham stimulation.
  Interventions: Procedure: Electrical stimulation
- Conditioning electrical stimulation (Experimental): Patients in the stimulation group will receive surgery as well as 1 hour of 20 Hz electrical stimulation 7 days prior to surgery
  Interventions: Procedure: Electrical stimulation

INTERVENTIONS:
Procedure: Electrical stimulation — Patients with cubital tunnel syndrome will receive either surgery and sham stimulation, or conditioning electrical stimulation 7 days prior to surgery

SUMMARY:
Cubital tunnel syndrome is the second most common compression neuropathy. In severe cases, functional recovery, even with surgery, is often poor. Therefore, alternative adjunct treatments capable of increasing the speed of nerve regeneration are much needed.

DETAILED DESCRIPTION:
The effect of brief conditioning electrical stimulation on nerve regeneration has been showed to be efficacy in animal studies. In this double-blind, randomized, controlled study, the investigators will compare the physiological and functional improvements post surgery compared with the controls who received surgery alone. Because electrical stimulation is reasonably well-tolerated and the treatment only takes an hour, it is a potentially feasible clinical tool for patients with severe nerve injury.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged >18 yr,
2. If signs and symptoms of severe CuTS (ie, McGowan-Goldberg grade 3) were observed,
3. If needle EMG examination showed evidence of chronic motor axonal loss and reduced recruitment in the ulnar-innervated intrinsic hand muscles, and
4. If electrophysiologic evidence of severe motor axonal loss with motor unit number estimation (MUNE) greater than 2 standard deviations below the normative mean.

Exclusion Criteria:

1) Patients were excluded if they had concurrent nerve injury, prior surgery for CuTS or coexisting neurologic conditions

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-06-28 (Estimated)

PRIMARY OUTCOMES:
Motor unit number estimation | 3 years
  A quantitative physiological measure of the number of motor nerve fibres in the target muscle

SECONDARY OUTCOMES:
Key pinch strength | 3 years
  A functional measure of the ulnar intrinsic hand muscles using a dynamometer
Disability of the Arm, Shoulder and Hand (DASH) Questionnaire | 3 years
  A questionnaire to quantify the severity of motor and sensory symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No